CLINICAL TRIAL: NCT04934137
Title: Development of Technologies to Increase In-Seat Movement to Prevent Sitting-Acquired Pressure Injuries in Wheelchair Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Minnesota (Other); Georgia Institute of Technology (Other)
Responsible Party: Principal Investigator, Susan Hallbeck, Ph.D., Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 19-008916; R01AG056255 (NIH)
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Pressure Ulcer; Pressure Injury; Wheelchair
Keywords: Pressure Injury; Pressure Ulcer; Weight Shift; Wheelchair; Pressure monitoring; Pressure relief
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensoria first intervention (Active Comparator): Group 1 participants will receive the Sensoria intervention during the first intervention phase for 4 weeks, and then the AW-Shift intervention during the second intervention phase for 4 weeks.
  Interventions: Behavioral: Sensoria; Behavioral: AW-Shift
- AW-Shift first intervention (Active Comparator): Group 2 participants will receive the AW-Shift intervention during the first intervention phase for 4 weeks, and then the Sensoria intervention during the second intervention phase for 4 weeks.
  Interventions: Behavioral: Sensoria; Behavioral: AW-Shift

INTERVENTIONS:
Behavioral: Sensoria — The Sensoria system uses a force-sensing mat installed under the wheelchair cushion that connects via Bluetooth to a mobile app. The mobile app displays information about weight shifts, goal-setting functions, and feedback on performance/outcomes.
Behavioral: AW-Shift — The AW-Shift system uses a pressure-sensing mat installed on top of the wheelchair cushion that connects via Bluetooth to a mobile app. The mobile app displays visual representation of the seating surface and can set reminders for weight shifts.

SUMMARY:
Pressure-related injuries in individuals with SCI and persons who use wheelchairs are one of the most dangerous secondary health problems encountered throughout the lifespan. With recurrence rates as high as 79% and mortality rates as high as 48% when sepsis is present, there exists a critical clinical need to target prevention of pressure injuries.

This study will examine the effects of two novel seat mapping technologies ("AW-Shift" and "Sensoria") on increasing in-seat movement in persons who may be at risk for pressure injuries due to altered sensation on their sitting surface. AW-Shift provides a visual display about pressure distribution directly between the body and the seat cushion to a wheelchair user outside of a clinical setting. Sensoria represents a novel technology to promote tissue health by providing users with information about their daily in-seat movement and providing weight shift reminders that are based on time since previous weight shift activities. Changes in the frequency of in-seat movement behaviors will be compared between baseline and each intervention period.

DETAILED DESCRIPTION:
For almost 50 years, clinicians and researchers have been interested in devices to monitor pressure and weight shift frequency, send alerts, provide cues, or track movement patterns in wheelchair users.

Despite the prevention efforts implemented over the years, pressure injuries continue to occur at a high rate of incidence. Without sensation to guide the need for changes in position to alleviate pressure, individuals with decreased sensation move significantly less than individuals with normal sensory systems. Thus, movement is a potentially robust protective factor to target. When focusing on movement as a modifiable risk factor, there is evidence that more in-seat movement is protective in wheelchair users. Behaviors, such as weight shifting to relieve pressure, decay over time, which could be attributed to lack of sensation to provide a natural cue to move. More work is needed to understand the types of movement that are most beneficial, and how to empower wheelchair users to move more often.

Our hypotheses are that A) Individuals will complete more frequent and more consistent weight shifts with access to the feedback systems compared to baseline and B) Self-efficacy beliefs for completing weight shifts will increase with use of the feedback systems.

This study will examine the effects of two novel seat mapping technologies ("AW-Shift" and "WiSAT") on increasing in-seat movement in persons who may be at risk for pressure injuries due to altered sensation on their sitting surface. AW-Shift provides a rich visual display about pressure distribution directly between the body and the seat cushion to a wheelchair user outside of a clinical setting. WiSAT represents a novel technology to promote tissue health by providing users with information about their daily in-seat movement and providing weight shift reminders that are based on time since previous weight shift activities. Changes in the frequency of in-seat movement behaviors will be compared between baseline and each intervention period.

The successful completion of this project will make large advancements in optimizing feedback about pressure and movement that will help wheelchair users become more effective in managing pressure distribution on an ongoing, daily basis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Be able to come to Mayo Clinic, UMN, or Georgia Tech campuses for study visits, or participate in virtual video study visits;
* Use a skin protection and positioning wheelchair cushion;
* Be able to perform weight shifts independently without assistance of another person (by moving themselves or using of power tilt);
* Own and are able to operate a smartphone with Apple or Android operating system;
* Are willing to download and use the mobile apps on their phone

Exclusion Criteria:

* Are scheduled for flap surgery;
* There is an active stage 3, 4, or unstageable pressure injury as defined by the National Pressure Injury Advisory Panel definitions anywhere on their sitting surface at time of enrollment;
* Use of a custom molded wheelchair cushion or alternating air cushion;
* Have/use the recline function on their manual or power wheelchair;
* Have a prescribed or limited sitting time of less than 5 hours per day;
* Live in a long-term care facility or group home and require 24 hours/day assistance;
* Have a known history of any condition or factor judged by the investigator to preclude participation in the study or which might hinder adherence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hallbeck, PhD, Principal Investigator — Mayo Clinic; Tamara Vos-Draper, PhD, OT, Principal Investigator — University of Minnesota; Sharon Sonenblum, PhD, Principal Investigator — Georgia Institute of Technology; Melissa Morrow, PhD, Principal Investigator — University of Texas
Locations (4):
- United States (4):
  - Georgia Institute of Technology, Atlanta, Georgia
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Texas Medical Branch, Galveston, Texas

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sensoria First Intervention | AW-Shift First Intervention
Started (Includes only participants who completed the baseline data collection, prior to intervention periods.) | 23 (Includes participants who completed the baseline data collection, prior to intervention periods.) | 23 (Includes participants who completed the baseline data collection, prior to intervention periods.)
Completed Baseline and Both Interventions (Includes participants who completed at least baseline and 2 intervention periods. This milestone should occur time-wise after the "Completed" milestone, but for analysis purposes it has been added as clarifying information per the comments. Participants who completed baseline and at least 1 intervention period are included as "Completed" and were analyzed.) | 15 (Includes participants who completed at least baseline and 2 intervention periods. Please note some participants in this group completed both interventions, and some did not due to time constraints, or intervention may not have been appropriate for all participants. We analyzed participants who completed baseline and at least 1 intervention who also had usable data.) | 14 (Includes participants who completed at least baseline and 2 intervention periods. Please note some participants in this group completed both interventions, and some did not due to time constraints, or intervention may not have been appropriate for all participants. We analyzed participants who completed baseline and at least 1 intervention who also had usable data.)
Completed (Includes participants who completed at least baseline and 1 intervention period.) | 21 (Includes participants who completed at least baseline and 1 intervention period. Please note some participants in this group completed both interventions, and some did not due to time constraints, or intervention may not have been appropriate for all participants. We analyzed participants who completed baseline and at least 1 intervention who also had usable data.) | 20 (Includes participants who completed at least baseline and 1 intervention period. Please note some participants in this group completed both interventions, and some did not due to time constraints, or intervention may not have been appropriate for all participants. We analyzed participants who completed baseline and at least 1 intervention who also had usable data.)
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Population: Includes participants who completed baseline collection and at least 1 intervention who had usable data to analyze. Some participants were not appropriate for both interventions and may have only completed 1 intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sensoria First Intervention | AW-Shift First Intervention | Total
Number analyzed (Participants) | 18 | 12 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 12 | 26
  >=65 years | 4 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.83 (14.21) | 42.92 (12.00) | 46.47 (13.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 10 | 6 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 15 | 11 | 26
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 12 | 30

OUTCOME MEASURES:

1. Primary Outcome: Normalized Weight Shift Frequency (Weight Shifts/Hour)
Description: The normalized average weight shift frequency per hour of wheelchair occupancy for each intervention phase. For each day of the intervention phases, a total number of weight shifts are measured per day in each phase. The total number of weight shifts are normalized by dividing by the number of hours of wheelchair occupancy for each day. Then finally, for each phase, the normalized average weight shift frequency is calculated by averaging across the daily normalized weight shift frequency for each phase.
Time Frame: The outcome measure was assessed at week 4 (the end) of each intervention period.
Population: Analysis population for each arm includes participants who had usable data who completed that intervention, regardless of which was completed first. Some participants completed both interventions and will be included in both "arms". Some participants were not appropriate for both interventions and only completed 1, but were still included in analysis because they had usable data and completed at least 1 intervention period.
Measure: Mean (Standard Deviation); unit: normalized weight shifts per hour
Groups:
- Participants Who Completed Sensoria Intervention: Group 1 participants will receive the Sensoria intervention during 4 weeks of the study. This includes all participants who used Sensoria regardless of which intervention they used first.
  Sensoria: The Sensoria system uses a force-sensing mat installed under the wheelchair cushion that connects via Bluetooth to a mobile app. The mobile app displays information about weight shifts, goal-setting functions, and feedback on performance/outcomes.
- Participants Who Completed AW-Shift Intervention: Group 2 participants will receive the AW-Shift intervention during 4 weeks of the study. This includes all participants who used AW-Shift regardless of which intervention they used first.
  AW-Shift: The AW-Shift system uses a pressure-sensing mat installed on top of the wheelchair cushion that connects via Bluetooth to a mobile app. The mobile app displays visual representation of the seating surface and can set reminders for weight shifts.
Arm/Group | Participants Who Completed Sensoria Intervention | Participants Who Completed AW-Shift Intervention
Number analyzed (Participants) | 27 | 18
normalized weight shifts per hour | 2.41 (1.93) | 2.38 (2.03)

ADVERSE EVENTS:
Time Frame: Adverse events were collected before and after each intervention phase at approximately 2, 6, and 12 weeks after the start of the baseline phase of the study.
Description: Participants at Risk for AE reporting cannot be provided for each intervention separately. Pts are allocated to each arm based on which intervention they completed first. However, some pts did not complete both interventions due to shortened timelines, drop out, or due to one of the interventions not being appropriate for the pt. We have analyzed all pts who completed baseline and 1 intervention who had usable data. Some of these participants completed both interventions, and some only 1.
Arm/Group | Sensoria First Intervention | AW-Shift First Intervention
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/12
Other Adverse Events (participants affected / at risk) | 0/18 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT04934137/Prot_SAP_001.pdf